Item number: 2022JC046

Jilin Province Health Science and Technology Capacity Improvement

**Project Task Book** 

Project Leader Category: Key Laboratory (Key Specialty)

Discipline: Internal Medicine of Traditional Chinese Medicine

Project Title: Study on the proteomics effect of Chuanhong stroke capsule

on patients with acute cerebral infarction

Applicant: Ding Yingyue

Undertaking unit: Changchun University of Traditional Chinese Medicine

Application Date: 27.4.2023

Jilin Provincial Health Commission

## **Informed Consent - Consent Signature Page**

Name of clinical research project: Study on the effect of Chuanhong Zhongfeng Capsule on proteomics of patients with acute cerebral infarction

**Unit in charge of the project:** The Affiliated Hospital of Changchun University of Traditional Chinese Medicine

## **Consent Statement:**

I have read the above description of this study and have had the opportunity to discuss and ask questions about this study with my physician, and my questions have been answered to my satisfaction.

I am aware of the possible benefits and inconveniences of participating in this study, I understand that participation is voluntary, and I confirm that I have had sufficient time to consider this and understand that:

- 1. I can ask my doctor for more information at any time;
- 2. I can withdraw from this study at any time without receiving discrimination or retaliation, and that my medical treatment and rights will not be affected.

I also understand that I need to cooperate with the investigator to record the changes in my condition and related information, and to complete the corresponding physical examination and biological sample retention during my participation in the study, which will be very beneficial to the improvement of my condition and the smooth implementation of the whole study.

I agree that the Ethics Committee or the representative of the investigator from the Affiliated Hospital of Changchun University of Traditional Chinese Medicine may have access to my study data.

Finally, I have decided to agree to participate in this study and to follow the researcher's arrangements as much as possible.

## **Patient Signature:**

Patient's contact phone number:

Date

## **Investigator Statement:**

I confirm that the details of this study have been explained to the patient, including his/her rights and obligations, as well as the possible benefits and

inconveniences, and that a copy of the signed informed consent form has been kept by the patient.

**Investigator's Signature:** 

**Investigator's work phone number:** 

Date